CLINICAL TRIAL: NCT00482222
Title: A Prospective Randomised Open Label Trial of Oxaliplatin/Fluoropyrimidine Versus Oxaliplatin/Fluoropyrimidine Plus Cetuximab Pre and Post Operatively in Patients With Resectable Colorectal Liver Metastasis Requiring Chemotherapy
Brief Title: Combination Chemotherapy With or Without Cetuximab Before and After Surgery in Treating Patients With Resectable Liver Metastases Caused By Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southampton (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000549541; USCTU-4351; USCTU-EPOC; EUDRACT-2006-003121-82; ISRCTN22944367; EU-20732
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2008-04

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: adenocarcinoma of the colon; stage IV colon cancer; adenocarcinoma of the rectum; stage IV rectal cancer; liver metastases; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Capecitabine; Fluorouracil; Leucovorin; Oxaliplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OxMdG / IrMdG chemotherapy (Active Comparator): OxMdG / IrMdG chemotherapy for 12 weeks Followed by surgery OxMdG / IrMdG chemotherapy for 12 weeks
  Interventions: Drug: capecitabine; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Other: study of socioeconomic and demographic variables; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: quality-of-life assessment
- OxMdG / IrMdG chemotherapy with cetuximab (Experimental): OxMdG / IrMdG chemotherapy with cetuximab for 12 weeks Followed by Surgery OxMdG / IrMdG chemotherapy with cetuximab for 12 weeks
  Interventions: Biological: cetuximab; Drug: capecitabine; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Other: study of socioeconomic and demographic variables; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: quality-of-life assessment

INTERVENTIONS:
Biological: cetuximab
  Arms: OxMdG / IrMdG chemotherapy with cetuximab
Drug: capecitabine
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Other: study of socioeconomic and demographic variables
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, fluorouracil, leucovorin, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving combination chemotherapy together with monoclonal antibodies before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery. It is not yet known whether combination chemotherapy is more effective with or without cetuximab in treating liver metastases caused by colorectal cancer.

PURPOSE: This randomized phase III trial is studying combination chemotherapy to compare how well it works when given with or without cetuximab before and after surgery in treating patients with resectable liver metastases caused by colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare progression-free survival of patients with resectable colorectal liver metastases treated with neoadjuvant and adjuvant combination chemotherapy with vs without cetuximab.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Compare the cost effectiveness of these regimens in these patients.

OUTLINE: This is a prospective, randomized, multicenter, open-label study. Patients are stratified according to participating center and assigned chemotherapy regimen. Patients are randomized to 1 of 2 treatment arms.

* Neoadjuvant therapy:

  * Arm I: Patients receive 1 of the following chemotherapy regimens:

    * OxMdG: Patients receive leucovorin calcium IV over 2 hours and oxaliplatin IV over 2 hours on day 1. Patients also receive fluorouracil IV continuously over 46 hours beginning on day 1. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
    * CAPOX: Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive 1 of the following regimens:

    * OxMdG + cetuximab: Patients receive cetuximab IV over 1-2 hours on day 1 and OxMdG chemotherapy as in arm I. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
    * CAPOX + cetuximab: Patients receive cetuximab IV over 1-2 hours on days 1, 8, and 15 and CAPOX chemotherapy as in arm I. Treatment repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Surgery: Beginning 2-6 weeks after completion of chemotherapy, patients in both arms undergo liver resection.
* Adjuvant therapy: Beginning 4-8 weeks after completion of surgery, patients receive treatment (OxMdG or CAPOX with or without cetuximab) as in arm I or II of neoadjuvant therapy.

  * Arm I: Treatment with OxMdG repeats every 2 weeks for up to 6 courses and treatment with CAPOX repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Treatment with OxMdG + cetuximab repeats every 2 weeks for up to 6 courses and treatment with CAPOX + cetuximab repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 12 weeks during chemotherapy, at completion of study treatment, every 3 months for 1 year, and then every 6 months thereafter.

Cost per life year and per quality-adjusted life year is assessed at baseline, every 12 weeks during treatment, and then at 3, 5, and 10 years.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* or radiologically confirmed primary adenocarcinoma of the colon or rectum

  * Advanced and/or metastatic disease NOTE: *Liver metastases should not be biopsied
* Must have potentially resectable liver metastases present, as defined by any of the following:

  * Metachronous metastases AND complete resection of the primary tumor without gross or microscopic evidence of residual disease (R0)
  * Synchronous metastases AND R0 resection of the primary tumor > 1 month before study entry
  * Synchronous metastases with sufficient evidence (e.g., by CT scan or diagnostic laparoscopy) that both the primary tumor and the liver metastases can be completely resected during the same procedure and resection of primary tumor can be delayed for 3-4 months
  * Suboptimally resectable disease (i.e., potentially resectable disease with compromise of the resection margins)
* No detectable extrahepatic tumor that cannot be completely resected
* Unidimensionally measurable disease
* No brain metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* WBC ≥ 4,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count > 150,000/mm³
* Bilirubin ≤ 1.25 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* AST or ALT ≤ 3 times ULN
* Creatinine clearance > 50 mL/min OR glomerular filtration rate > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No psychiatric or neurological condition that would preclude study compliance
* No partial or complete bowel obstruction
* No preexisting neuropathy > grade 1
* No other prior or concurrent malignant disease that, in the opinion of the investigator, would preclude study treatment
* No concurrent severe uncontrolled medical illness (including poorly-controlled angina or myocardial infarction within the past 3 months) that would preclude study treatment
* No known hypersensitivity reaction to any of the components of the study drugs

PRIOR CONCURRENT THERAPY:

* No prior systemic chemotherapy for metastatic disease
* More than 6 months since prior adjuvant chemotherapy comprising fluorouracil, leucovorin calcium, capecitabine, or irinotecan hydrochloride
* More than 1 month since prior rectal chemoradiotherapy comprising fluorouracil and leucovorin calcium
* No concurrent contraindicated medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2007-02; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | end of study

SECONDARY OUTCOMES:
Response rate before surgery as assessed by RECIST criteria | end of study
Pathological resection status | end of study
Overall survival | end of study
Toxicity | end of study
Quality of life as assessed by the EQ-5D, EORTC QLQ-C30, and EORTC QLQ-LMC21 | end of study
Cost effectiveness | end of study
Safety | end of study

CONTACTS AND LOCATIONS:
Overall Officials: John N. Primrose, MD, Study Chair — University Hospital Southampton NHS Foundation Trust
Locations (22):
- United Kingdom (22):
  - Basildon University Hospital, Basildon, England
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Addenbrooke's Hospital, Cambridge, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Aintree University Hospital, Liverpool, England
  - Royal Liverpool University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - UCL Cancer Institute, London, England
  - Royal Marsden - London, London, England
  - Charing Cross Hospital, London, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - St. Mary's Hospital, Newport, England
  - Cancer Research Centre at Weston Park Hospital, Nottingham, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Salisbury District Hospital, Salisbury, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Worthing Hospital, Worthing, England
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - University Hospital of Wales, Cardiff, Wales